CLINICAL TRIAL: NCT03216343
Title: Efficacy and Safety of Chiauranib in Relapsed/Refractory Small Cell Lung Cancer: a Single-arm, Open-label, Multi-center, Exploratory Phase Ib Study
Brief Title: Phase Ib/II Study of Chiauranib in Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR105
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — chiauranib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Patients take Chiauranib capsules 50mg, orally once daily, 28 days as a cycle until objective disease progression
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — CS2164

SUMMARY:
Chiauranib , which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

Because of its broad preclinical anti-tumor efficacy and the potential to improve conventional TKI kinase inhibitor therapy in various cancer indications,Chiauranib has now entered phase Ib clinical trials.

This clinical trial is studying the efficacy and safety of chiauranib works in treating patients with relapsed or refractory small cell lung cancer, in the meantime, exploreing the latent biomarkers accompany with chiauranib, as well as the relevancy of which and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤75 years;
2. Cytologically or histologically confirmed small cell lung cancer;
3. Patients have received at least 2 different systemic chemotherapy regimens (contained platinum based regimen) , and progressed or relapsed
4. At least one measurable lesion that can be accurately assessed ( RECIST1.1 criteria). If the only site of measurable disease is in a previously irradiated area, the patient must have documented progression of disease in this area.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Laboratory criteria are as follows:

   Complete blood count: hemoglobin (Hb) ≥80g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets >=75×109/L Biochemistry test: total bilirubin≦1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≦2.5×ULN(ALT,AST≦5×ULN if liver involved); serum creatinine(cr)≦1.5×ULN; Coagulation test: International Normalized Ratio (INR) < 1.5.
7. Life expectancy of at least 12 weeks.
8. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Patients receiving any anti-cancer therapy (including chemotherapy, target therapy, immunotherapy, radiotherapy, and anti-cancer Chinese traditional medicine, et al) within 4 weeks from the last dose prior to study entry; Subjects receiving any supportive treatment for haematology (including transfusion, blood products, or drugs that stimulate blood cells growth like G-CSF, et al) within 2 weeks from the last dose prior to study entry;
2. Patients with second primary cancer, except: adequately treated basal cell or squamous cell skin cancer, curatively treated in-situ cancer of the cervix, unless received curative treatment and with documented evidence of no recurrence during the past five years;
3. Patients with uncontrolled or significant cardiovascular disease, including:

   A) Grade II or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (NYHA Classification) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage.

   B) Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al).

   C) History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male),QTc≥470ms（female）at screening.

   D) Symptomatic coronary heart disease requiring treatment. E) Uncontrolled hypertension (> 140/90 mmHg) with single medication.
4. History of active bleeding within 6 months prior to screening; or patients receiving anticoagulation therapy; or patients with upper GI bleeding potential; or patients with active hemoptysis.
5. Patients with uncontrolled pleural effusion, pericardial effusion or ascites.
6. Patients with untreated central nervous system (CNS) metastasis; or requiring corticosteroids, anticonvulsants for CNS diseases treatment; or with evidence of progression or haemorrhage within 1 month prior to study entry; or clinical evidence of brain stem or leptomeninx involvement.
7. History of deep vein thrombosis or pulmonary embolism.
8. History of interstitial lung disease(ILD).
9. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
10. Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc), or undergone gastrectomy. .
11. 6 weeks or less from the last major surgery that involved general anaesthesia, or 2 weeks or less from the last minor surgery prior to screening (excluding placement of vascular access ) .
12. Proteinuria positive(≥1g/24h).
13. Patients with active or unable to control infections including human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, or other serious infectious diseases.
14. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study;
15. Any previous treatment with aurora kinase inhibitors, or VEGF/VEGFR inhibitors.
16. Candidates with drug and alcohol abuse.
17. Women of childbearing potential not willing to use and utilize an adequate method of contraception (such as intrauterine device, contraceptive and condom) throughout treatment and for at least 12 weeks after the last dose; pregnant or breastfeeding women; the result of urine pregnancy test was positive at screening; Man participants not willing to use and utilize an adequate method of contraception throughout treatment.
18. Any other condition which is inappropriate for the study according to investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate(ORR) | Up to a minimum 24 weeks after the last participant's first dose, or progression, or 75% subjects died.
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Number of subjects with Adverse Events as a Measure of Safety and Tolerability | Up to a minimum 28 weeks after the last participant's first dose, or progression, or 75% subjects died.
  Safety evaluation as measured by adverse events (AE), vital signs，electrocardiograph(ECG) and abnormal laboratory results according to CTCAE V4.03
Disease-control rate (DCR) | Up to a minimum 24 weeks after the last participant's first dose, or progression, or 75% subjects died.
Time to progression(TTP) | From date of the first dose of study drug until the date of first documented progression NOT including death, assessed up to 24 months
Duration of response (DOR) | from the date of first documented objective response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Progression-free survival (PFS) | From date of the first dose of study drug until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall survival (OS) | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months

OTHER OUTCOMES:
Median score of immunohistochemical expressed by Aurora B、CSF-1R and Myc protein. | assessed up to 24 months
Screening characteristics of ctDNA measurement (single gene analysis). | assessed up to 24 months
Screening characteristics of ctDNA measurement (multi-gene analysis). | assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No